CLINICAL TRIAL: NCT00260819
Title: Effects of Bosentan (Tracleer) in the Course of Pulmonary Artery Hypertension Induced by Hypoxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle Brindel, Department Clinical Research of Developpement
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P050502; AOR05038
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2007-03

CONDITIONS: Hypoxia-Induced Pulmonary Artery Hypertension
Keywords: Hypoxia-induced pulmonary artery hypertension; High-altitude pulmonary oedema; ETA receptor antagonist
MeSH Terms: conditions — Altitude Sickness | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Experimental and Placebo Comparator administered in random order during to successive experimental phase
  Interventions: Drug: Bosentan
- 2 (Placebo Comparator): Experimental and Placebo Comparator administered in random order during to successive experimental phase
  Interventions: Drug: Bosentam TRACLEER

INTERVENTIONS:
Drug: Bosentan — Single dose administration of 250 mg bosentan (2 pills Tracleer 125 mg) or placebo
  Other Names: TRACLEER
  Arms: 1
Drug: Bosentam TRACLEER — Single dose administration of 250 mg bosentan (2 pills Tracleer 125 mg) or placebo
  Arms: 2

SUMMARY:
Excessive rise in pulmonary artery pressure induced by low oxygen tension (hypoxia) is one of the factors implicated in high-altitude pulmonary oedema. Plasma ET1 increases in subjects exposed to high altitude and is correlated to pulmonary artery pressure.

The aim of the study is to investigate whether blockade of ET1 receptors would reduce the acute rise in systolic pulmonary artery pressure induced by hypoxia.

DETAILED DESCRIPTION:
Patients will be examined on a variable load supine bicycle ergometer. The exercise table will be tilted laterally by 20 to 30 degrees to the left. PASP will be assessed using Doppler echocardiography at rest and during during supine bicycle exercise in NORMOXIA and hypoxia. Exposure to normobaric hypoxia will be performed by breathing a hypoxic gas mixture at sea level during 90 minutes (12,3 % O2 + 87.7 % N2) reproducing conditions at 4300 m altitude. Exercise will be started at an initial workload of 40 watts and increased by 10 watts every minute to reach a workload level defined by a heart rate (HR) corresponding to 50% of the estimated maximal aerobic power

ELIGIBILITY:
Inclusion Criteria:

* 20 non smoker healthy volunteers : 10 resistant to high-altitude pulmonary oedema and 10 susceptible subjects, without history of cardiac or pulmonary disease or asthma, after a complete clinical examination and safety laboratory measurements prior to randomization, and after giving informed written consent.

Exclusion Criteria:

* antecedent of lung disease notably with asthmatic antecedent or HTAP
* antecedent of heart disease
* female genital organ
* systolic blood pressure < 85 mmHg or > 160 mmHg after 5 minutes of lengthened rest.
* sentimentality in a medicine, in particular in a bosentan or in one of the excipients of the tablet.
* hepatic incapacity moderated to severe correspondent in the class B or C of the classification of Child-Pugh (cf Pharmacokinetics) Rate serous hepatic aminotransferases, aspartate aminotransferases( ASAT) and\or alanine aminotransférases ( ALAT), superior to 3 times the superior limit of the normal before the started of the treatment.
* pointed or chronic systematic diseases.
* presence of antibody anti-HIV, of anti-HVC antibody, antigens Hbs and\or antibody anti-Hbc. - active addiction to smoking.
* alcohol abuse and of toxins.
* Taking of concomitant medicines except those allowed the chapter concomitant treatments.
* signs, symptoms or values of the biological examinations situated except the clinically acceptable values for healthy subjects with or without antecedent of OPHA.
* common(current) ingestion of excessive quantities of tea, coffee(cafe), chocolate and\or drinks containing some caffeine (> 5 cups / day, is approximately 500 mg of caffeine a day).
* consumption of juice of grapefruit and\or herb tea on base of St.
* John's wort
* Don of blood in 3 months preceding the study.
* Persons in period of exclusion on the national file of the persons lending itself to the biomedical search(research) without direct individual profit.
* refusal or linguistic or psychic incapacity to sign the lit(enlightened) assent.
* subject which can not submit itself to the constraints of the protocol (for example, not cooperative, incapable to go(surrender) to the visits of follow-up and probably incapable to finish the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To investigate whether bosentan compared to placebo reduces hypoxia-induced increase in pulmonary artery pressure in healthy subjects and in subjects with past history of high-altitude pulmonary oedema | during the study

SECONDARY OUTCOMES:
To compare | during the study
pulmonary artery pressure response to exercise, | during the study
exercise capacity, | during the study
oxygen desaturation, | during the study
and to assess the global safety | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Michel AZIZI, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre d'Investigation Clinique 9201 Hôpital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Result] Grunig E, Mereles D, Hildebrandt W, Swenson ER, Kubler W, Kuecherer H, Bartsch P. Stress Doppler echocardiography for identification of susceptibility to high altitude pulmonary edema. J Am Coll Cardiol. 2000 Mar 15;35(4):980-7. doi: 10.1016/s0735-1097(99)00633-6. PMID 10732898